CLINICAL TRIAL: NCT01239381
Title: Phase II Study of Individualized Stereotactic Body Radiotherapy of Liver Metastases
Brief Title: Individualized Stereotactic Body Radiotherapy of Liver Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hannah Roberts, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-139; Other (Other Grant/Funding Number: program income earned on C06 CA059267)
Record Dates: First submitted 2010-06-14; First posted 2010-11-11 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor; Liver Metastases
Keywords: proton radiation; stereotactic body radiotherapy; SBRT

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SBRT-Proton (Experimental): Stereotactic body radiotherapy by proton radiation
  Interventions: Radiation: Stereotactic body radiotherapy-proton

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy-proton — Dose will be determined by the size and location of the tumor(s); 2-3 treatments per week for two weeks

SUMMARY:
Stereotactic body radiation therapy (SBRT) is a technique that is used to deliver radiation, to sites in the body. All participants in this study will be treated with SBRT using proton beam radiation. Proton beam radiation uses tiny particles to deliver radiation to tumors. The purpose of this research study is to determine if SBRT with protons will prevent tumor growth and reduce the treatment side effects for liver metastases.

DETAILED DESCRIPTION:
* Participants receiving SBRT with protons, will receive radiation treatment as an outpatient at the Francis H. Burr Proton Therapy Center at Massachusetts General Hospital.
* Not everyone who participates in this study will be receiving the same dose of radiation. The dose received will be determined by the size and location of the tumor(s).
* Participants will receive 2-3 SBRT treatments per week for two weeks.
* During radiation therapy visits the following tests/procedures will be performed: vital signs, physical examination, routine blood tests, research blood tests, and radiation planning.
* Follow-up assessments will be performed once at 9 weeks after study treatment, then at 6 months, 12 months, 18 months and 24 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven cancer diagnosis of a solid tumor with 1-4 liver metastases. There is no upper size limit. Liver metastases may be diagnosed by imaging alone, no liver biopsy is required. Extrahepatic disease is allowed if it have been stable for 3 months prior to study entry, the dominant disease burden is intrahepatic and the patient is referred for definitive radiation therapy to the disease in the liver
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension as 10mm or greater with spiral CT scan
* Patients may have had prior chemotherapy, targeted biological therapy, surgery, transarterial chemoembolization (TACE), radiofrequency ablation, or cryosurgery for their disease as long as the prior therapy occured greater than 3 weeks elapsed before the first radiation treatment. Patients may not have had prior liver directed radiation, including radioembolization.
* 18 years of age or older
* Expected survival must be greater than three months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Patients must have at least 800mL of uninvolved liver
* Normal organ and marrow function as outlined in the protocol
* If patient has underlying cirrhosis, only Child-Pugh classification Group A patients should be included in this study. Clinical assessment of ascites and encephalopathy is required. Child-Pugh classification must be determined for all study participants at the time of eligibility analysis.
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation

Exclusion Criteria:

* Women who are pregnant or lactating
* Patients with gross ascites or encephalopathy
* Local conditions or systemic illnesses which would reduce the local tolerance to radiation treatment, such as serious local injuries, active collagen vascular disease, etc.
* Prior liver directed radiation treatment, including selective internal radiation
* No serious medical illness, which may limit survival to less than 3 months
* No serious psychiatric illness which would limit compliance with treatment
* Participants who have had chemotherapy or radiotherapy within 3 weeks prior to starting study treatment or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier
* Participants may not be receiving any other investigational agents, or any other anti-cancer therapy during treatment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia.
* Only solid tumors are permitted. Thus, individuals with a liver mass from a diagnosis of lymphoma or leukemia are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2010-10-05 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2017-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hannah J. Roberts, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institue, Boston, Massachusetts

REFERENCES:
- [Derived] Hong TS, Wo JY, Borger DR, Yeap BY, McDonnell EI, Willers H, Blaszkowsky LS, Kwak EL, Allen JN, Clark JW, Tanguturi S, Goyal L, Murphy JE, Wolfgang JA, Drapek LC, Arellano RS, Mamon HJ, Mullen JT, Tanabe KK, Ferrone CR, Ryan DP, Iafrate AJ, DeLaney TF, Zhu AX. Phase II Study of Proton-Based Stereotactic Body Radiation Therapy for Liver Metastases: Importance of Tumor Genotype. J Natl Cancer Inst. 2017 Sep 1;109(9). doi: 10.1093/jnci/djx031. PMID 28954285

RESULTS

PARTICIPANT FLOW:
Groups:
- SBRT-Proton: Stereotactic Body Radiation Therapy (SBRT) by proton radiation
  Stereotactic body radiotherapy-proton: Dose will be determined by the size and location of the tumor(s); 2-3 treatments per week for two weeks
Period: Overall Study
Arm/Group | SBRT-Proton
Started | 92
Completed | 90
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Patients that were registered but did not start study therapy were not included in the analysis.
Groups:
- SBRT-Proton: SBRT by proton radiation
  Stereotactic body radiotherapy-proton: Dose will be determined by the size and location of the tumor(s); 2-3 treatments per week for two weeks
Arm/Group | SBRT-Proton
Number analyzed (Participants) | 90
Age, Continuous [Median (Full Range); unit: years] | 68 [34 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 57
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 90
Primary Cancer Site [Count of Participants; unit: Participants]
  Colorectal | 35
  Pancreatic | 16
  Esophagogastric | 12
  Hepatocellular | 8
  Lung | 5
  Gallbladder | 3
  Breast | 3
  Small Bowel or Duodenal | 3
  Anal | 2
  Head and Neck | 2
  Prostate | 1
Number of Tumors [Count of Participants; unit: Participants]
  1 Tumor | 54
  2 Tumors | 21
  3 Tumors | 10
  4 Tumors | 5
Median Tumor Size [Median (Full Range); unit: Centimeters (cm)] — Median Tumor size among the 142 tumors analyzed
  Centimeters (cm) | 2.55 [0.48 to 11.9]
Categorical Tumor size [Count of Participants; unit: Participants] — Population: 88 participants with complete tumor size data
  Participants
    ≤ 5 cm: number analyzed (Participants) | 88
    ≤ 5 cm | 50
    > 5 cm: number analyzed (Participants) | 88
    > 5 cm | 31
    > 10 cm: number analyzed (Participants) | 88
    > 10 cm | 7

OUTCOME MEASURES:

1. Primary Outcome: Local Control Rate
Description: The percentage of participants with local control at primary tumor site at one year. Local is evaluated using Response Evaluation Criteria In Solid Tumors (RECIST). Local control is defined as achieving either Complete response (CR), Partial Response (PR), or Stable Disease (SD).
  * (CR): Disappearance of entire lesion, with no additional evidence of disease.
  * (PR): At least a 30% decrease in the (sum of) the longest diameter (LD) of the primary lesion, taken as reference the baseline sum LD.
  * (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: 1 year
Population: The 90 participants that started study treatment
Measure: Number; unit: percentage of participants
Arm/Group | SBRT-Proton
Number analyzed (Participants) | 90
percentage of participants | 77

2. Secondary Outcome: Median Follow-up Time
Description: The median follow-up time among the 39 participants still alive at the time of analysis, measured from the start of treatment until the time of analysis.
Time Frame: 1 year
Population: the 39 participants still alive at the time of analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | SBRT-Proton
Number analyzed (Participants) | 39
Months | 11 [0.3 to 41]

3. Secondary Outcome: Median Overall Survival
Description: The median overall survival (in months) of participants as measured from the start of treatment.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | SBRT-Proton
Number analyzed (Participants) | 90
Months | 18 [14 to 21]

4. Secondary Outcome: Median Progression Free Survival
Description: The median amount of time participants survived without cancer progression following the start of study treatment. Progression was assessed using RECIST v1.0. Progressive Disease (PD) is defined as at least a 20% increase in the Longest Diameter (LD) of the lesion, taken as the reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 1 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | SBRT-Proton
Number analyzed (Participants) | 90
Months | 4 [3 to 8]

5. Secondary Outcome: 2-year Local Control Rate
Description: The percentage of participants with local control 2 years after the start of study treatment.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SBRT-Proton
Number analyzed (Participants) | 90
percentage of participants | 65.8 [55.8 to 75.6]

6. Secondary Outcome: 1 Year Local Control Rate Among Participants With Colorectal Cancer
Description: The percentage of participants with local control at one year among the participants with colorectal cancer as the primary cancer.
Time Frame: 1 year
Population: Participants with colorectal cancer
Measure: Number; unit: percentage of participants
Arm/Group | SBRT-Proton
Number analyzed (Participants) | 35
percentage of participants | 60

7. Secondary Outcome: Median Survival Among Participants With Colorectal Cancer
Description: The median amount of time participants survived from the start of treatment, among the participants with colorectal cancer.
Time Frame: 2 years
Population: The 35 participants with colorectal cancer as the primary cancer.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | SBRT-Proton
Number analyzed (Participants) | 35
Months | 18 [13 to 32]

ADVERSE EVENTS:
Time Frame: From the start of treatment until 30 days after the completion of treatment
Description: Participants are assessed for adverse events twice during treatment, after 4 weeks of followup, and then every three months until 24 months post treatment.
Arm/Group | SBRT-Proton
All-Cause Mortality (participants affected / at risk) | 1/90
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 86/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBRT-Proton (N=90)
Ear pain (Ear and labyrinth disorders) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 10 (22)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 3 (3)
Palpitations (Cardiac disorders) | 1 (4)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Chills (General disorders) | 2 (3)
Edema limbs (General disorders) | 7 (16)
Fatigue (General disorders) | 70 (205)
Fever (General disorders) | 4 (4)
Gait disturbance (General disorders) | 2 (3)
Localized edema (General disorders) | 1 (1)
Malaise (General disorders) | 3 (7)
Non-cardiac chest pain (General disorders) | 3 (7)
Pain (General disorders) | 15 (28)
General disorders and administration site conditions - Other, (General disorders) | 2 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5 (18)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (4)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 5 (8)
Abdominal distension (Gastrointestinal disorders) | 3 (6)
Abdominal pain (Gastrointestinal disorders) | 35 (90)
Ascites (Gastrointestinal disorders) | 2 (4)
Bloating (Gastrointestinal disorders) | 7 (12)
Constipation (Gastrointestinal disorders) | 10 (16)
Diarrhea (Gastrointestinal disorders) | 14 (30)
Dyspepsia (Gastrointestinal disorders) | 5 (8)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (5)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (6)
Gastroparesis (Gastrointestinal disorders) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 22 (34)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 4 (6)
Stomach pain (Gastrointestinal disorders) | 1 (3)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (8)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 5 (7)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (2)
Rash pustular (Infections and infestations) | 1 (2)
Upper respiratory infection (Infections and infestations) | 5 (11)
Urinary tract infection (Infections and infestations) | 4 (4)
Infections and infestations - Other, specify (Infections and infestations) | 3 (6)
Bruising (Injury, poisoning and procedural complications) | 5 (14)
Dermatitis radiation (Injury, poisoning and procedural complications) | 40 (101)
Fall (Injury, poisoning and procedural complications) | 2 (3)
Fracture (Injury, poisoning and procedural complications) | 1 (5)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 10 (19)
Alkaline phosphatase increased (Investigations) | 12 (33)
Aspartate aminotransferase increased (Investigations) | 10 (20)
Blood bilirubin increased (Investigations) | 8 (25)
Blood prolactin abnormal (Investigations) | 1 (2)
Lymphocyte count decreased (Investigations) | 2 (5)
Platelet count decreased (Investigations) | 5 (16)
Serum amylase increased (Investigations) | 1 (1)
Weight gain (Investigations) | 5 (11)
Weight loss (Investigations) | 8 (14)
White blood cell decreased (Investigations) | 2 (3)
Investigations - Other, specify (Investigations) | 5 (10)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 25 (49)
Dehydration (Metabolism and nutrition disorders) | 2 (6)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (24)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 4 (7)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (8)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (26)
Musculoskeletal and connective tissue disorder - (Musculoskeletal and connective tissue disorders) | 4 (6)
Akathisia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 9 (11)
Dysgeusia (Nervous system disorders) | 1 (3)
Headache (Nervous system disorders) | 4 (6)
Memory impairment (Nervous system disorders) | 4 (4)
Paresthesia (Nervous system disorders) | 2 (4)
Peripheral motor neuropathy (Nervous system disorders) | 2 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (10)
Somnolence (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Eye pain (Eye disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 5 (8)
Confusion (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 6 (13)
Insomnia (Psychiatric disorders) | 6 (7)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (14)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (3)
Proteinuria (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (4)
Urinary incontinence (Renal and urinary disorders) | 1 (3)
Urinary retention (Renal and urinary disorders) | 1 (2)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 3 (8)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (3)
Flushing (Vascular disorders) | 1 (1)
Hematoma (Vascular disorders) | 2 (2)
Hot flashes (Vascular disorders) | 2 (3)
Hypertension (Vascular disorders) | 4 (6)
Superficial thrombophlebitis (Vascular disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes